CLINICAL TRIAL: NCT02185365
Title: Evaluation of T1rho Magnetic Resonance Imaging for Diagnosis of Cartilage Lesions in Hips With Developmental Dysplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Zimmer Biomet (Industry); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20140371-01H
Record Dates: First submitted 2014-06-02; First posted 2014-07-09 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Developmental Dysplasia of the Hip
Keywords: T1-rho MRI; dGEMRIC MRI; DDH; Developmental dysplasia of the hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Developmental dysplasia of the hip (DDH): Patients will complete 2 magnetic resonance imaging (MRI): T1-rho and dGEMRIC. The T1-rho MRI does not require the injection of a contrast agent, while the dGEMRIC MRI requires a gadolinium injection to visualize cartilage in the hip.
  Interventions: Radiation: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging (MRI) — Patients will undergo 2 different MRIs of the affected hip. Both MRIs assess hip cartilage degeneration. A contrast agent, Gadolinium, will be used to visualize cartilage during the MRI. The contrast agent is injected through an intravenous (a small plastic tube inserted into a vein in the patients' arm) before the MRI.

SUMMARY:
One of the leading causes of hip arthritis is developmental dysplasia of the hip (DDH). DDH can lead to major damage in the hip joint and may result in hip arthritis later in life. Patients recruited into this study will be undergoing corrective hip surgery within the next 6 months with a goal of preventing further hip problems down the road. This study is being done to see how well a newer type of Magnetic Resonance Imaging (MRI) detects hip cartilage damage compared to an older but well validated MRI method.

DETAILED DESCRIPTION:
The start of arthritis can first be detected in certain molecules in the joint. Proteoglycan is a molecule that is important to cartilage structure, and is lost as arthritis develops. Magnetic resonance imaging (MRI) is one of the best ways to image cartilage, and an investigational MRI technique that has shown great promise in detecting proteoglycan amounts is called T1-rho.

In this study, patients with hip dysplasia will undergo this investigational MRI in addition to a well validated MRI method (called dGEMRIC) to see if T1-rho is as good as dGEMRIC at detecting cartilage damage. The dGEMRIC MRI requires an injection of a contrast agent, while the T1-rho MRI does not. If the T1-rho is shown to be as useful as the dGEMRIC method it can then be used to look at cartilage damage in the hip without having to have an injection.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of developmental dysplasia of the hip (DDH)

Exclusion Criteria:

* patients under the age of 18
* pregnancy and/or lactation
* non-MRI compatible implants (stents, electronic devices, cardiac pacers or wires)
* severe claustrophobia
* prior contrast allergic reaction
* kidney impairment
* previous hip surgery
* osteoarthritis on conventional radiographs (Tönnis Grade>0)
* additional underlying hip diseases such as posttraumatic arthritis, Legg-Calvé-Perthes-Disease (LCPD), or slipped capital femoral epiphysis (SCFE)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will consist of patients diagnosed with developmental dysplasia of the hip (DDH), and who are scheduled to undergo surgery to correct this.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Assess proteoglycan amounts in hip cartilage | Within the 6 months prior to surgery
  Our aim is to correlate T1-rho with dGEMRIC values in painful hips with underlying DDH. To achieve this, we will assess whether T1-rho MRI values correlate with dGEMRIC MRI values in hips with DDH.

SECONDARY OUTCOMES:
Change in WOMAC Questionnaire | 12 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is widely used as a standard assessment of arthritis in the hip joint. The Index is self-administered and assesses the three dimensions of pain (5 items), joint stiffness (2 items), and Physical Function (17 items) in hip osteoarthritis using 24 questions. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme. These correspond to an ordinal scale of 0-4. Scores are summed with higher scores indicating worse pain, stiffness, and function.
Change in iHOT 12 Questionnaire | 12 months
  The International Hip Outcome Tool (iHOT-12) is a questionnaire that has recently been validated in young active patients with early hip disease. The questionnaire is self-administered and assesses across 4 domains: symptoms and functional limitations; sport and recreational activities; job-related concerns; and social, emotional, and lifestyle concerns. Questions are answered by marking a visual analog scale between 2 anchor statements (100-mm scale). The total score is calculated as a simple mean of these responses ranging from 0 to 100, with 100 representing the best possible quality-of-life score.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beaule, MD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No